CLINICAL TRIAL: NCT04278313
Title: Randomized Controlled Trial of Ovarian Function Following Intraovarian Injection of Platelet Rich Plasma for Women With Ovarian Aging
Brief Title: Ovarian Function Following Intraovarian Injection of PRP
Acronym: PRP4POA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Center for Human Reproduction (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 02102020-0
Record Dates: First submitted 2020-02-18; First posted 2020-02-20 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Diminished Ovarian Reserve; Diminished Ovarian Reserve Due to Advanced Maternal Age
Keywords: Infertility - Ovarian dysfunuction; Diminished Ovarian Reserve; Premature Ovarian Aging (POA)

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to treatment with either Platelet Rich Plasma (PRP) or Platelet Poor Plasma (PPP)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRP group (Experimental): Platelet RICH Plasma prepared using RegenLab FDA approved device.
  Interventions: Procedure: PRP - Platelet Rich Plasma
- PPP group (Placebo Comparator): Platelet POOR Plasma prepared using RegenLab FDA approved device.
  Interventions: Procedure: PPP - Platelet Poor Plasma

INTERVENTIONS:
Procedure: PRP - Platelet Rich Plasma — Using a sterile vacutainer technique two 8 ml samples of whole blood is drawn into two Regen Lab A-PRP vacutainers with gel separator and citrate. Invert the tube to mix with citrate. The whole blood undergoes two centrifugations, once for 3 minutes and again for 5 minutes. Using a 20-gauge 6-inch spinal needle 2 ml of Platelet POOR Plasma will be drawn off the supernatant from each tube to leave 2.5 ml of Platelet Rich Plasma in the tube. The tube is inverted several times to suspend the platelet pellet. The prepared plasma labeled with the participants name and randomization code will be transported to the procedure room.
  Arms: PRP group
Procedure: PPP - Platelet Poor Plasma — Using a sterile vacutainer technique two 8 ml samples of whole blood is drawn into two Regen Lab A-PRP vacutainers with gel separator and citrate. Invert the tube to mix with citrate. The whole blood undergoes two centrifugations, once for 3 minutes and again for 5 minutes. Using a 20-gauge 6-inch spinal needle 2 ml of Platelet POOR Plasma will be drawn off the supernatant from each tube. The prepared plasma will be transported to the procedure room. The prepared plasma labeled with the participants name and randomization code will be transported to the procedure room.
  Arms: PPP group

SUMMARY:
Consenting women with evidence of poor ovarian reserve will be randomly assigned to treatment with either Platelet Rich Plasma (PRP) or Platelet Poor Plasma (PPP).

DETAILED DESCRIPTION:
As women age oocytes are gradually depleted with a consequent progressive loss of ovarian function and fertility. When a woman's follicle cohort falls below a critical level, she enters a transitional time of diminished ovarian reserve known as ovarian aging. Recently the use of autologous platelet-rich plasma (A-PRP) has been proposed as an additional strategy for improving ovarian function. A-PRP is prepared from autologous blood using an FDA approved device. The rationale for the use of PRP is that it contains growth factors which stimulate cellular anabolism, inflammatory modulators that create an anti-inflammatory effect and fibrinogen which acts as a scaffold for regenerating tissue. The investigators hypothesize that the growth factors present in PRP may have a beneficial effect promoting growth and recruitment of antral follicles. The investigators will recruit a prospective cohort of 90 patients with evidence of Premature Ovarian Aging/DOR. Women invited to participate in this RCT will have FSH above 12 and AMH below 1.0 ng/mL respectively and will have had fewer than 6 oocytes retrieved in a previous ovulation attempt. Consenting participants in this trial will be randomized in a doubly blind fashion to two groups. One will receive Platelet Rich Plasma (PRP) and the other will receive Platelet Poor Plasma (PPP). Women assigned to PPP will be offerred PRP in a future cycle if they so desire.

ELIGIBILITY:
Inclusion Criteria:

* fewer than 6 oocytes in response to past ovulation induction
* desire to establish a pregnancy using IVF
* Age 44 years and under.
* FSH > 12
* AMH < 1.0
* No Aspirin or Motrin for one week before treatment

Exclusion Criteria:

* Age > 45 years
* Marked thrombocytopenia
* Blood diseases
* Hypofibrinogenemia
* Hemodynamic instability
* Anticoagulant or antiaggregant treatment
* Oncological diseases (specially, skeletal system and blood)
* Sepsis
* Acute and chronic infectious diseases
* Autoimmune diseases, for example, lupus erythematosus, etc.

Ages: 21 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Must have ovaries and desire to establish a pregnancy using IVF
Enrollment: 90 (Estimated)
Dates: Start 2020-02-24 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Embryo Transfer | 6 weeks
  Number of participants with at least one day-3 embryo 8-cell with less than 5% fragmentation in an IVF cycle

SECONDARY OUTCOMES:
Embryos Produced | 6 weeks
  Mean number of day-3 embryo 8-cell with less than 5% fragmentation produced
AMH | 4 weeks
  Serum concentration of Anti Mullerian Hormone
Antral Follicle Count | 4 weeks
  Number of Antral Follicles determined by pelvic sonogram on day 2 or 3 of menses

OTHER OUTCOMES:
Pregnancy | 8 weeks
  Number of patients who Establish a Clinical Pregnancy (Fetal pole and positive evidence of fetal heart on pelvic sonogram)

CONTACTS AND LOCATIONS:
Overall Officials: David H Barad, MD, Principal Investigator — Center for Human Reproduction
Locations (1):
- Center for Human Reproduction, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD